CLINICAL TRIAL: NCT02104362
Title: A Phase I-II Study to Evaluate Exclusive Single-fraction Irradiation by Interstitial High Dose Rate Brachytherapy in Patients With Prostate Cancer at Low Risk or at Low Intermediate Risk of Local Recurrence
Brief Title: Single Fraction Early Prostate Irradiation (SiFEPI)
Acronym: SiFEPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-A01514-41; 2013/16 (Other: Centre Antoine Lacassagne)
Record Dates: First submitted 2014-03-31; First posted 2014-04-04 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- exclusive single-fraction irradiation (Other)
  Interventions: Radiation: exclusive single-fraction irradiation

INTERVENTIONS:
Radiation: exclusive single-fraction irradiation

SUMMARY:
Recently, HDR brachytherapy delivering only a 19 Gy fraction was proposed as exclusive treatment for low and intermediate risk prostate cancers. With a median 3-year follow-up, the Spanish team reported a biochemical control rate of 100% and 87%, respectively, for low risk and intermediate risk tumors. In parallel with these encouraging results regarding biochemical control, the authors described excellent urinary and digestive tolerance, notably the absence of grade > 2 complications. However, it should be noted, in this study, that special protection was provided to the anterior aspect of the rectum by means of a 10 ml transperineal injection of hyaluronic acid into the prostate-rectal interspace.

The idea of using a single high dose (in one fraction) was proposed at the MSKCC by the team of Fucks et al. which, in 2008, following a median 18-month follow-up, published a a 90% local control rate for spinal metastases after a single dose at 18 to 24 Gy.

The aim of the present study is to analyze acute urinary and digestive toxicity (< 180 days) observed following interstitial high dose rate prostate brachytherapy delivering a total dose of 20 Gy in one fraction.

DETAILED DESCRIPTION:
Expected benefit(s) of the trial

* Improved quality of life during brachytherapy on account of the absence of radioactive seeds in the prostate:

  * Fewer early urinary complications,
  * No urine filtration,
  * No post-operative use of condoms,
  * No 2-year ban on cremation following treatment,
* Health cost savings,
* Acquisition of dosimetric data for inverse optimization.

Predictable risk(s) for patients Predictable risks in the context of this trial involve the frequency of essentially urinary disorders.

Methodology Open, monocentric, phase I-II study.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from histologically-proven adenocarcinoma-type prostate cancer:

  * with low risk of biochemical recurrence
  * with a low intermediate risk of biochemical recurrence (maximum of 1 intermediate risk factor)*
  * stage T1c, T2a, T2b
  * Gleason score 6 (3+3) or 7 (3+4) with at most 3 positive biopsies
* PSA < 15 ng/ml
* Age ≥ 18 years
* Karnofsky index ≥ 70%
* Life expectancy ≥ 10 years
* No contraindication to injection of hyaluronic acid in the prostate-rectal interspace
* Patient aware of the information leaflet and having signed the informed consent form
* Patient covered by medical insurance

Exclusion Criteria:

* Stage ≥ T2c
* Gleason score 7 (4+3) or ≥ 8
* PSA > 15 ng/ml
* Presence of the following anatomico-pathological criteria:

  * Involvement of the nerve fibers
  * Peri-tumoral vascular embolisms
  * Capsule involvement
  * Number of positive biopsies ≥ 50%
  * 100% positive biopsies in a lobe
  * Involvement of the seminal vesicle
* Prostate volume ≥60 cc
* Large prostatic transurethral resection and/or dating from less than 6 months
* Poor urinary function in the absence of alpha-blockers

  * IPSS score > 15
  * Post-mictional residue > 50 cc
  * Flow rate with Qmax < 12 ml/s
* Remote metastasis
* Neoadjuvant anti-androgenic treatment
* Prior treatment with pelvic irradiation and/or chemotherapy
* Active infection or other underlying severe pathology likely to prevent the patient from receiving treatment
* History of cancer other than basocellular cutaneous cancer or other form of cancer in complete remission for more than 5 years
* Evolving psychiatric disorder
* Vulnerable persons as defined by article L1121-5 to -8

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
acute urinary toxicity occurring within 6 months after irradiation. | up to 5 years
  to assess the acute urinary toxicity occurring within 6 months after irradiation.

SECONDARY OUTCOMES:
acute digestive toxicity occurring during the 6 months following irradiation | up to 5 years
  Assessment of acute digestive toxicity occurring during the 6 months following irradiation,

OTHER OUTCOMES:
Local recurrence-free survival at 5 years | up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Antoine Lacassagne, Nice, France

REFERENCES:
- See also: Related Info — http://www.centreantoinelacassagne.org